CLINICAL TRIAL: NCT01208675
Title: The Swedish BioFINDER Study: Early Diagnosis of Alzheimer's Disease - a Multidisciplinary Approach
Brief Title: The Swedish BioFINDER Study
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Erik Stomrud, M.D., PhD, Skane University Hospital
Other Study IDs: TiDiS-2010
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Dementia With Lewy Bodies; Vascular Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, plasma, DNA, mRNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild cognitive impairment: 550 patients with mild cognitive impairment or subjective cognitive symptoms at baseline.
- Healthy elderly subjects: 650 elderly subjects, who are cognitively healthy at baseline.

SUMMARY:
The present study aims at combining biochemical methods with various types of imaging techniques to identify the pathophysiology of Alzheimer's disease (AD). The main interest is to find markers associated with the very early steps in the pathology of this disease. The investigators shall thus screen for i) molecules in cerebrospinal fluid (CSF) and plasma specific for AD, and ii) brain imaging markers (e.g. MRI and PET) that correlate to detailed clinical assessments.

Biomarkers of interest would then be useful to:

1. Enable accurate detection of the disease early on. Such biomarkers need to specifically reflect the very early pathophysiology of AD and distinguish it from disorders with similar symptomatology, such as other types of dementia and major depression. The sensitivity and specificity of these biomarkers in combination with clinical assessment should be of at least 90%.
2. Enable prediction of the course of events of the disease, such as the disease rate in individual patients. Biomarkers that can predict the pattern of future symptoms will be extremely valuable.
3. Allow monitoring of early effects of new disease-modifying therapies (so-called surrogate biomarkers). Currently clinical therapeutic trials for AD require large patient groups together with long-term treatment. Both size of the groups and treatment time will be reduced with the help of surrogate biomarkers.
4. Study the pathogenesis of the disease. Biomarkers can be used to investigate in detail early alterations in AD patients. For instance, changes in the levels of certain molecules in CSF together with genetic predisposition could then be correlated to clinical signs and changes detectable by brain imaging. This can lead to identification of new therapeutic targets that could easily be monitored in future trials.

DETAILED DESCRIPTION:
1. Baseline investigations of patients with mild cognitive deficits

   We are conducting a prospective, longitudinal study in which we consecutively include patients with mild cognitive deficits (MCI), who seek medical care at the Neuropsychiatric Clinic (Malmö, Sweden) or Unit for Cognitive Medicine (Lund, Sweden). At baseline the MCI patients undergo detailed neurological and psychiatric examination, including assessment of depressive symptoms and ADL-capacity as well as cognitive and motor tests. Patients are also genotyped for APOE. Samples of plasma, blood (for DNA and mRNA) and CSF are also collected. All patients undergo an advanced MRI scan of the brain. A subset will undergo 18F-Flutemetamol PET. We will include patients over a period of three years.

   1.2 Follow-up of MCI patients

   Thereafter, we follow patients for up to 10 years with repeated testing and clinical evaluation. During clinical follow-up we estimate how many of the patients develop any type of dementia, for instance AD. Moreover we also estimate how aggressive the progression of the disease is in those patients that develop AD with the help of repeated cognitive testing.
2. Baseline investigations of healthy elderly volunteers

   To answer the question if new biomarkers could detect early signs of AD in healthy people, we have included cognitively healthy elderly subjects. These people are recruited from a population-based study in Malmö ("Malmö Kost Cancer") where people without memory problems or cognitive difficulties, and who performs well on cognitive tests, are offered to participate. These individuals will undergo the same baseline studies that MCI patients (see above), including cognitive tests, psychiatric assessment, lumbar puncture, blood tests and MRI scan. A subset is also examined with 18F-Flutemetamol PET.

   2.1 Follow-up of elderly volunteers

   This population will also be followed-up for 10 years with repeated cognitive tests to determine which subjects develop cognitive impairment (e.g. memory problems) over this period of time.
3. Analyses of CSF and plasma/blood

   CSF and plasma/blood sampling is done at baseline, 2, 4, 6 and 10 years of follow-up. To find novel and better biomarkers to predict AD in both healthy and MCI patients, the CSF, plasma and blood will be analyzed by various biomedical techniques. We will also screen for biomarkers that can help us to predict how fast the disease will progress. We will use two different approaches, namely: a) analysis of various candidate biomarkers and b) unbiased screening using proteomics.
4. Magnetic resonance imaging (MRI) MRI is done at baseline, 2, 4 and 6 years of follow-up, using the same MRI scanner. We will evaluate the potential benefits of new MRI protocols for prediction of future AD. MRI will also be used to study the pathogenesis of AD. These new approaches include: 3D-MP RAGE, T2* GRE, DTI/DTT, ASL and MRS.

ELIGIBILITY:
Inclusion Criteria:

Healthy elderly subjects

* No cognitive symptoms reported by patient and/or informant
* Normal performance on cognitive tests
* General cognition and functional performance preserved such that a diagnosis of MCI or dementia cannot be made by physician at the time of the baseline visit
* Between 60 and 90 years of age
* Fluent in Swedish
* Agrees to at least one lumbar puncture, and neuropsychological testing.

Mild cognitive impairment

* Cognitive symptoms reported by patient and/or informant
* Between 60 and 80 years of age
* Mini-Mental State Exam score between 24 and 30
* General cognition and functional performance sufficiently preserved such that a diagnosis of dementia cannot be made by physician at the time of the baseline visit
* Fluent in Swedish
* Agrees to at least one lumbar puncture, and neuropsychological testing.

Exclusion Criteria (for both MCI and healthy elderly):

* Any significant neurologic disease other than dementia disorders, such as Huntington's disease, normal pressure hydrocephalus, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
* Major depression as described in DSM-IV.
* History of schizophrenia or other recurrent psychotic disorder
* History of alcohol or substance abuse or dependence within the past 5 years

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
To compare the time to conversion to clinically probable AD in MCI subjects or healthy elderly subjects with normal and abnormal biomarkers (CSF, blood, MRI, PET) | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 4-6 years after baseline.

SECONDARY OUTCOMES:
Rate of cognitive decline as measured by various cognitive tests, Activities of Daily Living (FAQ) and Global Deterioration Scale. | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 10 years after baseline.
Group differences for imaging and wet biomarker measurements. | At baseline, 1 years, 2 years, 3 years, 4 years, 6 years, 8 years and 10 years.
Rate of volume change of structural MRI measures and amyloid PET | At baseline, 1 years, 2 years, 3 years, 4 years, 6 years, 8 years and 10 years.
Rates of change on each specified biochemical biomarker | At baseline, 1 years, 2 years, 3 years, 4 years, 6 years, 8 years and 10 years.
Correlations between biomarkers and biomarker change | At baseline, 1 years, 2 years, 3 years, 4 years, 6 years, 8 years and 10 years.
Subgroups analyses: Abnormal CSF biomarkers, positive amyloid imaging, APOE genotype. | At baseline, 1 years, 2 years, 3 years, 4 years, 6 years, 8 years and 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Hansson, MD, PhD, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Memory Clinic, Hospital of Ängelholm, Ängelholm
  - Memory Clinic, Skåne University Hospital, Malmo

REFERENCES:
- [Background] Hansson O, Janelidze S, Hall S, Magdalinou N, Lees AJ, Andreasson U, Norgren N, Linder J, Forsgren L, Constantinescu R, Zetterberg H, Blennow K; Swedish BioFINDER study. Blood-based NfL: A biomarker for differential diagnosis of parkinsonian disorder. Neurology. 2017 Mar 7;88(10):930-937. doi: 10.1212/WNL.0000000000003680. Epub 2017 Feb 8. PMID 28179466
- [Background] Janelidze S, Hertze J, Nagga K, Nilsson K, Nilsson C; Swedish BioFINDER Study Group; Wennstrom M, van Westen D, Blennow K, Zetterberg H, Hansson O. Increased blood-brain barrier permeability is associated with dementia and diabetes but not amyloid pathology or APOE genotype. Neurobiol Aging. 2017 Mar;51:104-112. doi: 10.1016/j.neurobiolaging.2016.11.017. Epub 2016 Dec 5. PMID 28061383
- [Background] Smith R, Scholl M, Honer M, Nilsson CF, Englund E, Hansson O. Tau neuropathology correlates with FDG-PET, but not AV-1451-PET, in progressive supranuclear palsy. Acta Neuropathol. 2017 Jan;133(1):149-151. doi: 10.1007/s00401-016-1650-1. Epub 2016 Nov 29. No abstract available. PMID 27900460
- [Background] Mattsson N, Zetterberg H, Janelidze S, Insel PS, Andreasson U, Stomrud E, Palmqvist S, Baker D, Tan Hehir CA, Jeromin A, Hanlon D, Song L, Shaw LM, Trojanowski JQ, Weiner MW, Hansson O, Blennow K; ADNI Investigators. Plasma tau in Alzheimer disease. Neurology. 2016 Oct 25;87(17):1827-1835. doi: 10.1212/WNL.0000000000003246. Epub 2016 Sep 30. PMID 27694257
- [Background] Hahn A, Schain M, Erlandsson M, Sjolin P, James GM, Strandberg OT, Hagerstrom D, Lanzenberger R, Jogi J, Olsson TG, Smith R, Hansson O. Modeling Strategies for Quantification of In Vivo 18F-AV-1451 Binding in Patients with Tau Pathology. J Nucl Med. 2017 Apr;58(4):623-631. doi: 10.2967/jnumed.116.174508. Epub 2016 Oct 20. PMID 27765859
- [Background] Smith R, Schain M, Nilsson C, Strandberg O, Olsson T, Hagerstrom D, Jogi J, Borroni E, Scholl M, Honer M, Hansson O. Increased basal ganglia binding of 18 F-AV-1451 in patients with progressive supranuclear palsy. Mov Disord. 2017 Jan;32(1):108-114. doi: 10.1002/mds.26813. Epub 2016 Oct 6. PMID 27709757
- [Background] Smith R, Puschmann A, Scholl M, Ohlsson T, van Swieten J, Honer M, Englund E, Hansson O. 18F-AV-1451 tau PET imaging correlates strongly with tau neuropathology in MAPT mutation carriers. Brain. 2016 Sep;139(Pt 9):2372-9. doi: 10.1093/brain/aww163. Epub 2016 Jun 29. PMID 27357347
- [Background] Surova Y, Lampinen B, Nilsson M, Latt J, Hall S, Widner H; Swedish BioFINDER study; van Westen D, Hansson O. Alterations of Diffusion Kurtosis and Neurite Density Measures in Deep Grey Matter and White Matter in Parkinson's Disease. PLoS One. 2016 Jun 30;11(6):e0157755. doi: 10.1371/journal.pone.0157755. eCollection 2016. PMID 27362763
- [Background] Pannee J, Portelius E, Minthon L, Gobom J, Andreasson U, Zetterberg H, Hansson O, Blennow K. Reference measurement procedure for CSF amyloid beta (Abeta)1-42 and the CSF Abeta1-42 /Abeta1-40 ratio - a cross-validation study against amyloid PET. J Neurochem. 2016 Nov;139(4):651-658. doi: 10.1111/jnc.13838. Epub 2016 Sep 30. PMID 27579672
- [Background] Janelidze S, Stomrud E, Palmqvist S, Zetterberg H, van Westen D, Jeromin A, Song L, Hanlon D, Tan Hehir CA, Baker D, Blennow K, Hansson O. Plasma beta-amyloid in Alzheimer's disease and vascular disease. Sci Rep. 2016 May 31;6:26801. doi: 10.1038/srep26801. PMID 27241045
- [Background] van Westen D, Lindqvist D, Blennow K, Minthon L, Nagga K, Stomrud E, Zetterberg H, Hansson O. Cerebral white matter lesions - associations with Abeta isoforms and amyloid PET. Sci Rep. 2016 Feb 9;6:20709. doi: 10.1038/srep20709. PMID 26856756
- [Background] Smith R, Wibom M, Olsson T, Hagerstrom D, Jogi J, Rabinovici GD, Hansson O. Posterior Accumulation of Tau and Concordant Hypometabolism in an Early-Onset Alzheimer's Disease Patient with Presenilin-1 Mutation. J Alzheimers Dis. 2016;51(2):339-43. doi: 10.3233/JAD-151004. PMID 26836192
- [Background] Hall S, Surova Y, Ohrfelt A; Swedish BioFINDER Study; Blennow K, Zetterberg H, Hansson O. Longitudinal Measurements of Cerebrospinal Fluid Biomarkers in Parkinson's Disease. Mov Disord. 2016 Jun;31(6):898-905. doi: 10.1002/mds.26578. Epub 2016 Feb 16. PMID 26878815
- [Background] Voevodskaya O, Sundgren PC, Strandberg O, Zetterberg H, Minthon L, Blennow K, Wahlund LO, Westman E, Hansson O; Swedish BioFINDER study group. Myo-inositol changes precede amyloid pathology and relate to APOE genotype in Alzheimer disease. Neurology. 2016 May 10;86(19):1754-61. doi: 10.1212/WNL.0000000000002672. Epub 2016 Apr 15. PMID 27164711
- [Background] Janelidze S, Zetterberg H, Mattsson N, Palmqvist S, Vanderstichele H, Lindberg O, van Westen D, Stomrud E, Minthon L, Blennow K; Swedish BioFINDER study group; Hansson O. CSF Abeta42/Abeta40 and Abeta42/Abeta38 ratios: better diagnostic markers of Alzheimer disease. Ann Clin Transl Neurol. 2016 Jan 1;3(3):154-65. doi: 10.1002/acn3.274. eCollection 2016 Mar. PMID 27042676
- [Background] Palmqvist S, Zetterberg H, Mattsson N, Johansson P; Alzheimer's Disease Neuroimaging Initiative; Minthon L, Blennow K, Olsson M, Hansson O; Swedish BioFINDER Study Group. Detailed comparison of amyloid PET and CSF biomarkers for identifying early Alzheimer disease. Neurology. 2015 Oct 6;85(14):1240-9. doi: 10.1212/WNL.0000000000001991. Epub 2015 Sep 9. PMID 26354982
- [Background] Lindqvist D, Prokopenko I, Londos E, Middleton L, Hansson O. Associations between TOMM40 Poly-T Repeat Variants and Dementia in Cases with Parkinsonism. J Parkinsons Dis. 2016;6(1):99-108. doi: 10.3233/JPD-150693. PMID 26756745
- [Background] Gustavsson AM, Stomrud E, Abul-Kasim K, Minthon L, Nilsson PM, Hansson O, Nagga K. Cerebral Microbleeds and White Matter Hyperintensities in Cognitively Healthy Elderly: A Cross-Sectional Cohort Study Evaluating the Effect of Arterial Stiffness. Cerebrovasc Dis Extra. 2015 May 20;5(2):41-51. doi: 10.1159/000377710. eCollection 2015 May-Aug. PMID 26120319
- [Background] Hall S, Surova Y, Ohrfelt A, Zetterberg H, Lindqvist D, Hansson O. CSF biomarkers and clinical progression of Parkinson disease. Neurology. 2015 Jan 6;84(1):57-63. doi: 10.1212/WNL.0000000000001098. Epub 2014 Nov 19. PMID 25411441
- [Background] Palmqvist S, Zetterberg H, Blennow K, Vestberg S, Andreasson U, Brooks DJ, Owenius R, Hagerstrom D, Wollmer P, Minthon L, Hansson O. Accuracy of brain amyloid detection in clinical practice using cerebrospinal fluid beta-amyloid 42: a cross-validation study against amyloid positron emission tomography. JAMA Neurol. 2014 Oct;71(10):1282-9. doi: 10.1001/jamaneurol.2014.1358. PMID 25155658
- [Background] Lautner R, Palmqvist S, Mattsson N, Andreasson U, Wallin A, Palsson E, Jakobsson J, Herukka SK, Owenius R, Olsson B, Hampel H, Rujescu D, Ewers M, Landen M, Minthon L, Blennow K, Zetterberg H, Hansson O; Alzheimer's Disease Neuroimaging Initiative. Apolipoprotein E genotype and the diagnostic accuracy of cerebrospinal fluid biomarkers for Alzheimer disease. JAMA Psychiatry. 2014 Oct;71(10):1183-91. doi: 10.1001/jamapsychiatry.2014.1060. PMID 25162367
- [Background] Silajdzic E, Constantinescu R, Holmberg B, Bjorkqvist M, Hansson O. Flt3 ligand does not differentiate between Parkinsonian disorders. Mov Disord. 2014 Sep;29(10):1319-22. doi: 10.1002/mds.25948. Epub 2014 Jul 16. PMID 25044107
- [Background] Lindqvist D, Hall S, Surova Y, Nielsen HM, Janelidze S, Brundin L, Hansson O. Cerebrospinal fluid inflammatory markers in Parkinson's disease--associations with depression, fatigue, and cognitive impairment. Brain Behav Immun. 2013 Oct;33:183-9. doi: 10.1016/j.bbi.2013.07.007. Epub 2013 Jul 31. PMID 23911592
- [Background] Surova Y, Szczepankiewicz F, Latt J, Nilsson M, Eriksson B, Leemans A, Hansson O, van Westen D, Nilsson C. Assessment of global and regional diffusion changes along white matter tracts in parkinsonian disorders by MR tractography. PLoS One. 2013 Jun 13;8(6):e66022. doi: 10.1371/journal.pone.0066022. Print 2013. PMID 23785466
- [Derived] Cullen NC, Leuzy A, Palmqvist S, Janelidze S, Stomrud E, Pesini P, Sarasa L, Allue JA, Proctor NK, Zetterberg H, Dage JL, Blennow K, Mattsson-Carlgren N, Hansson O. Individualized prognosis of cognitive decline and dementia in mild cognitive impairment based on plasma biomarker combinations. Nat Aging. 2021 Jan;1(1):114-123. doi: 10.1038/s43587-020-00003-5. Epub 2020 Nov 30. PMID 37117993
- [Derived] Johansson M, Stomrud E, Johansson PM, Svenningsson A, Palmqvist S, Janelidze S, van Westen D, Mattsson-Carlgren N, Hansson O. Development of Apathy, Anxiety, and Depression in Cognitively Unimpaired Older Adults: Effects of Alzheimer's Disease Pathology and Cognitive Decline. Biol Psychiatry. 2022 Jul 1;92(1):34-43. doi: 10.1016/j.biopsych.2022.01.012. Epub 2022 Jan 31. PMID 35346458